CLINICAL TRIAL: NCT00156182
Title: A Phase 2, Long-Term, Open-Label, Safety Extension Study of Asoprisnil (J867) in Patients With Uterine Leiomyomata
Brief Title: A Long-Term Safety Study of Asoprisnil in the Treatment of Uterine Fibroids.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M01-275
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2008-05

CONDITIONS: Leiomyoma
Keywords: Fibroid Uterus; Leiomyoma; Uterine Fibroids; asoprisnil
MeSH Terms: conditions — Leiomyoma | interventions — asoprisnil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil

INTERVENTIONS:
Drug: Asoprisnil — 10mg Tablet, oral Daily for 6 months

SUMMARY:
This study was designed to determine the long-term safety of asoprisnil 10 mg in women with one or more uterine fibroids after an initial 12 weeks in study M99-144.

DETAILED DESCRIPTION:
No medical therapy is currently available for the long-term treatment of uterine fibroids. The objective of this study is to determine the long-term safety of asoprisnil 10 mg daily for 6 months, after an initial 12 weeks in study M99-144, in women with one or more uterine fibroids, confirmed by ultrasound in study M99-144. The safety endpoints for this study will be based on ultrasound and endometrial biopsy results, adverse events, and any changes from baseline laboratory values and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Completed dosing and Day 84 procedures at sites in study M99-144
* No interruption of dosing
* Otherwise continued good health

Exclusion Criteria:

* Any abnormal lab result the study-doctor considers significant
* History of severe reaction to or current use of hormone therapy
* History of alcohol or drug abuse

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2001-04; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in uterine volume and volume of the largest fibroid from pre-treatment in study M99-144 | Treatment months 3 and 6 and Post-treatment months 3 and 6
Percentage of subjects that achieved amenorrhea. | Treatment months 1-6

SECONDARY OUTCOMES:
Improvement in hematologic parameters. | Treatment months 2,4,and 6
Improvement in Uterine fibroid symptoms(menorrhagia, metrorrhagia, pelvic pressure, bloating, urinary disorders, pelvic pain, dysmenorrhea, dyspareunia) using a 4 point scale | Treatment Months 1-6
Change from baseline in uterine size in gestational weeks. | Months 3 and 6
Duration of amenorrhea. | Start of previous study to first post-treatment menses.
Response to global efficacy question regarding improvement of fibroid symptoms. | Month 6
Mean change from baseline for endocrine determinations. | Months 2,4 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott